CLINICAL TRIAL: NCT01628068
Title: Efficacy of Left Atrial Appendage Closure After Gastrointestinal Bleeding
Brief Title: ELIGIBLE (Efficacy of Left atrIal Appendage Closure After GastroIntestinal BLEeding)
Acronym: ELIGIBLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Victoria Martin Yuste, MD, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELIGIBLE; Estudio ELIGIBLE (Other: Fundació Clínic)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Adverse Reaction to Drugs Affecting the Gastrointestinal System
Keywords: Left atrial appendage occlusion; gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left atrial appendage occlusion (Active Comparator): Left atrial appendage occlusion with Amplatzer device plus aspirine plus clopidogrel during 3 months
  Interventions: Device: Left atrial appendage occlusion
- Oral anticoagulation (No Intervention): Oral anticoagulation

INTERVENTIONS:
Device: Left atrial appendage occlusion — Left atrial appendage occlusion with Amplatzer device plus aspirine plus clopidogrel during 3 months
  Arms: Left atrial appendage occlusion

SUMMARY:
Patients with atrial fibrillation requiring anticoagulation treatment are at high risk of gastrointestinal bleeding. The investigators propose the percutaneous stop the oral anticoagulation and closure of the left atrial appendage with the Amplatzer ® system in patients receiving anticoagulant therapy for atrial fibrillation without associated valvular heart disease, to reduce significantly the risk of stroke while minimizing the risk of bleeding in a group of patients with high risk for both events.

ELIGIBLE trial(Left atrial appendage Efficacy of GastroIntestinal Bleeding after closure) is a prospective, multicentric and randomized (2 to 1) trial, comparing percutaneous closure of atrial appendage left versus standard treatment with oral anticoagulants in patients with history of gastrointestinal bleeding and high embolic risk.

ELIGIBILITY:
Inclusion Criteria:

* documented atrial fibrilation (paroxysmal or permanent) without significant heart valve disease
* > 18 years
* Classic oral anticoagulation(INR at therapeutic levels: 2-3) or New oral anticoagulants
* CHA2-DS2-VASC score ≥ 3
* prior digestive bleeding without any treatable cause
* Informed consent.

Exclusion Criteria:

* POF
* contraindication to further treatment with dual antiplatelet therapy (aspirin + clopidogrel)
* Intracardiac thrombus
* significant carotid disease
* Cardioversion scheduled within 30 days following the implantation
* AF not controlled by FVM> 100 bpm
* AF secondary to surgery or ablation
* thrombosis in patients <40 years
* chronic renal insufficiency with Cr clearance <30 ml 2
* left appendage sizeappendage with inlet <12.6 mm or > 28.5 (ETE)
* depth of the appendage <10mm in the TEE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Combined overall mortality, major bleeding, stroke or procedure-related complications | 1 year
  The primary end point will be at one year the combined overall mortality, major bleeding, stroke or procedure-related complications.
  1. Mortality from any cause
  2. Severe bleeding defined according to VARC criteria
  3. Ischemic stroke or hemorrhagic stroke at 12 months.
  4. Complications related to the procedure: include:
     * device embolization
     * severe pericardial effusion with hemodynamic compromise that requires drainage
     * Device thrombosis
     * cardiac perforation
     * major local complications (according to definitions of VARC)

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Infanta Cristina, Badajoz, Badajoz
  - Fundació Clínic per a la Recerca Biomèdica, Barcelona, Barcelona
  - Hospital de La Paz, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Mdrid
  - Hospital Virgen de la Victoria, Málaga, Málaga
  - Hospital Virgen de la Macarena, Seville, Sevilla